CLINICAL TRIAL: NCT02393430
Title: Clinical Effect of Rebamipide on Chronic Gastritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: BangMao Wang (Other)
Responsible Party: Sponsor-Investigator, BangMao Wang, Chief of Gastroenterology Department, Tianjin Medical University General Hospital
Organization: Tianjin Medical University General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GH 0123
Record Dates: First submitted 2014-11-23; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Gastritis
MeSH Terms: conditions — Gastritis | interventions — rebamipide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental (Experimental): The experimental group were treated with rebamipide 0.1g tid and optimization of life style.
  Interventions: Drug: Rebamipide; Behavioral: optimization of life style
- control (Placebo Comparator): The control group were only optimized their life style.
  Interventions: Behavioral: optimization of life style

INTERVENTIONS:
Drug: Rebamipide — Rebamipide is a
  Other Names: Mucosta
  Arms: experimental
Behavioral: optimization of life style

SUMMARY:
To investigate the clinical effect of rebamipide in chronic gastritis patients. Patients with chronic gastritis were randomly divided into the experimental group and the control group. The experimental group were treated with rebamipide 0.1g tid and optimization of life style, and the control group were only optimized their life style for 26 weeks. Upper gastrointestinal endoscopy was performed in all patients to evaluate the severity of gastritis by modified Lanza score (MLS) and the histology by the updated Sydney system before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* With the symptoms as follow: epigastric pain, abdominal discomfort, abdominal distention, poor appetite, nausea, vomiting and so on
* diagnosed as chronic gastritis with endoscopic and pathological methods
* agree to join in this clinical trail

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
modified Lanza score | 26 weeks
visual Analog scale | 26 weeks
  to describe the inflamamtory of gastric mucosa pathologically

CONTACTS AND LOCATIONS:
Overall Officials: Wang Bang-mao, Study Chair — Tianjin meidcal university general hospital,China